CLINICAL TRIAL: NCT02862730
Title: A Randomized, Four-way, Cross-over Outpatient Study to Assess the Efficacy of a Dual-hormone Versus Insulin Alone Closed-loop System With Exercise Detection vs a Predictive Low Glucose Suspend System vs Current Care
Brief Title: Four Way Crossover Closed Loop With Exercise Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jessica Castle, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15590
Record Dates: First submitted 2016-07-28; First posted 2016-08-11 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-08

CONDITIONS: Type 1 Diabetes
Keywords: diabetes; closed-loop; dual hormone; exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Predictive Low Glucose Suspend Arm (Experimental): Subjects will undergo an 84 hour study with 24 hours inpatient and 60 hour outpatient. The predictive low glucose suspend system will run through the artificial pancreas controller in predictive low glucose suspend mode and utilize the patient's optimized basal rates, correction factor, and carb ratio, but it will have the additional safety net of the pump suspending insulin when it predicts a hypoglycemic event.
  Interventions: Device: Artificial Pancreas Controller in Predictive Low Glucose Suspend Mode
- Dual Hormone Closed-loop Arm (Experimental): Subjects will undergo an 84 hour study with 24 hours inpatient and 60 hour outpatient using the closed-loop artificial pancreas controller in dual hormone mode to manage blood sugar that includes an exercise detection component that includes a reduction in insulin delivery and an increase in glucagon delivery upon detection.
  Interventions: Device: Artificial Pancreas Controller in Dual Hormone Mode
- Single Hormone Closed-loop Arm (Experimental): Subjects will undergo an 84 hour study with 24 hours inpatient and 60 hour outpatient using the closed-loop artificial pancreas controller in single hormone mode to manage blood sugar that includes an exercise detection component that includes a reduction in insulin delivery upon detection.
  Interventions: Device: Artificial Pancreas Controller in Single Hormone Mode
- Sensor Augmented Pump Therapy arm (Active Comparator): Subjects will undergo an 84 hour study with 24 hours inpatient and 60 hour outpatient with subject's insulin pump and glucose sensor, if he/she typically uses one. Subjects will still wear a heart rate monitor uploading to a smart phone.
  Interventions: Device: Subject's insulin pump

INTERVENTIONS:
Device: Artificial Pancreas Controller in Dual Hormone Mode — The artificial pancreas controller contains an algorithm for managing blood glucose in people with type 1 diabetes which includes an exercise detection component. The new algorithm will have 3 modes: a single hormone closed-loop insulin only mode, a dual-hormone closed-loop insulin and glucagon mode and an insulin only mode with predictive low glucose suspend. Closed-loop Artificial Pancreas Controller includes insulin and glucagon delivery algorithm implemented on a smart phone, utilizing sensor glucose values from a Dexcom G4 sensor and sending delivery commands to two Tandem t:slim insulin pumps, one filled with insulin and one with glucagon.
  Other Names: APC
  Arms: Dual Hormone Closed-loop Arm
Device: Subject's insulin pump — Subject will continue on their subcutaneous delivery of insulin on his/her own insulin pump using their own basal rates and carb ratios for meal boluses, managing their blood sugar as they normally would.
  Arms: Sensor Augmented Pump Therapy arm
Device: Artificial Pancreas Controller in Single Hormone Mode — The artificial pancreas controller contains an algorithm for managing blood glucose in people with type 1 diabetes which includes an exercise detection component. The new algorithm will have 3 modes: a single hormone closed-loop insulin only mode, a dual-hormone closed-loop insulin and glucagon mode and an insulin only mode with predictive low glucose suspend. Closed-loop Artificial Pancreas Controller includes insulin delivery algorithm implemented on a smart phone, utilizing sensor glucose values from a Dexcom G4 sensor and sending delivery commands to one Tandem t:slim insulin pumps filled with insulin.
  Arms: Single Hormone Closed-loop Arm
Device: Artificial Pancreas Controller in Predictive Low Glucose Suspend Mode — The artificial pancreas controller contains an algorithm for managing blood glucose in people with type 1 diabetes which includes an exercise detection component. The new algorithm will have 3 modes: a single hormone closed-loop insulin only mode, a dual-hormone closed-loop insulin and glucagon mode and an insulin only mode with predictive low glucose suspend. Closed-loop Artificial Pancreas Controller includes insulin delivery algorithm implemented on a smart phone, utilizing sensor glucose values from a Dexcom G4 sensor and sending delivery commands to one Tandem t:slim insulin pumps filled with insulin.
  Arms: Predictive Low Glucose Suspend Arm

SUMMARY:
Closed-loop systems are an emerging technology that automate hormone delivery. They are quickly paving the way to revolutionize the treatment of type 1 diabetes. Several categories have emerged: dual-hormone (insulin and glucagon) closed-loop systems and closed-loop systems with insulin only, one variety of which is the low glucose suspend safety feature now available from Medtronic (MiniMed 530G with Enlite). The study described within this protocol is designed to test the efficacy of a new closed-loop algorithm for managing blood glucose in people with type 1 diabetes before and after exercise. The new algorithm will have 3 modes: a single hormone insulin only mode, a dual-hormone insulin and glucagon mode and an insulin only mode with predictive low glucose suspend, all with an exercise detection algorithm. The purpose of this study is to determine whether a dual hormone AP with an exercise detection algorithm outperforms both single hormone AP and a low glucose suspend algorithm and sensor augmented pump therapy using the subject's own insulin pump.

DETAILED DESCRIPTION:
Subjects will undergo four approximately 84 hour studies. The first day of each study will be an approximately 12 hour inpatient visit to include activities of daily living and an exercise period with 2 days spent as an outpatient. The subject will come back to the research center on the fourth day to complete another approximately 12 hour inpatient visit to include activities of daily living and an exercise period followed by removal of all devices. In randomized order, subjects will have glucose controlled using the following systems: 1) dual-hormone closed-loop system, 2) insulin only closed-loop system, 3) predictive low glucose suspend system and 4) sensor augmented pump therapy with subject using their own insulin and insulin pump. Both of the closed-loop system algorithms have an exercise detection algorithm that uses inputs from a heart rate monitor and accelerometer, the Zephyrlife BioPatch. After exercise detection, insulin is turned off for the first 30 minutes, the total insulin infusion rate is adjusted by an exercise multiplier, and for the dual-hormone system, the target glucose for glucagon is increased along with the maximum dose of glucagon allowed. The predictive low glucose suspend system will utilize the patient's optimized basal rates, correction factor, and carb ratio. The patient will bolus for meals and hyperglycemia as usual under PLGS, but will have the additional safety net of the pump suspending insulin when it predicts a hypoglycemic event. The Dexcom CGM system and the Tandem t:slim pumps will be used for all three intervention visits.

Subjects will arrive at the CTRC at 7am at the start of intervention visits. Subjects will eat breakfast, lunch and dinner in the research center. Subjects will eat breakfast at 8:30am. After breakfast, subjects will complete activities of daily living (sitting on a chair, lying on a bed, washing dishes, sweeping the floor, etc.). Subjects will eat lunch at 12pm. Subjects will exercise for 45 minutes on a treadmill around 2pm. Subjects will eat dinner at 6pm and be discharged. The subject will then go home for Day 2 and Day 3 and return on Day 4 to complete another 12 hour inpatient visit with the schedule of activities identical to Day 1.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes mellitus for at least 1 year.
* Physically willing and able to perform 45 min of exercise (as determined by the investigator after reviewing the subjects activity level)
* Current use of an insulin pump.
* Lives with another person age 18 or older who will be present while subject exercises at home and that can attend the training on using the system with the subject.
* Lives within 20 miles of OHSU.
* A1C<10%
* Willingness to follow all study procedures, including attending all clinic visits.
* Willingness to sign informed consent and HIPAA documents.

Exclusion Criteria:

* Female of childbearing potential who is pregnant or intending to become pregnant or breast-feeding, or is not using adequate contraceptive methods. Acceptable contraception includes birth control pill / patch / vaginal ring, Depo-Provera, Norplant, an IUD, the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence.
* Any cardiovascular disease, defined as a clinically significant EKG abnormality at the time of screening or any history of: stroke, heart failure, myocardial infarction, angina pectoris, or coronary arterial bypass graft or angioplasty. Diagnosis of 2nd or 3rd degree heart block or any non-physiological arrhythmia judged by the investigator to be exclusionary.
* Renal insufficiency (GFR < 60 ml/min, using the MDRD equation as report by the OHSU laboratory).
* Liver failure, cirrhosis, or any other liver disease that compromises liver function as determined by the investigator.
* Hematocrit of less than or equal to 34%.
* Hypertensive subjects with systolic blood pressure >= 160 mmHg or diastolic blood pressure >= 100 mmHg despite treatment or who have treatment-refractory hypertension (e.g. requiring four or more medications).
* History of severe hypoglycemia during the past 12 months prior to screening visit or hypoglycemia unawareness as judged by the investigator. Subjects will complete a hypoglycemia awareness questionnaire. Subjects will be excluded for four or more R responses.
* Adrenal insufficiency.
* Any active infection.
* Known or suspected abuse of alcohol, narcotics, or illicit drugs.
* Seizure disorder.
* Active foot ulceration.
* Severe peripheral arterial disease characterized by ischemic rest pain or severe claudication.
* Major surgical operation within 30 days prior to screening.
* Use of an investigational drug within 30 days prior to screening.
* Chronic usage of any immunosuppressive medication (such as cyclosporine, azathioprine, sirolimus, or tacrolimus).
* Bleeding disorder, treatment with warfarin, or platelet count below 50,000.
* Allergy to aspart insulin.
* Allergy to glucagon.
* Insulin resistance requiring more than 200 units per day.
* Need for uninterrupted treatment of acetaminophen.
* Current administration of oral or parenteral corticosteroids.
* Any life threatening disease, including malignant neoplasms and medical history of malignant neoplasms within the past 5 years prior to screening (except basal and squamous cell skin cancer).
* Beta blockers or non-dihydropyridine calcium channel blockers.
* Current use of any medication intended to lower glucose other than insulin (ex. use of liraglutide).
* Diagnosis of pheochromocytoma, insulinoma, or glucagonoma, personal or family history of multiple endocrine neoplasia (MEN) 2A, MEN 2B, neurofibromatosis or von Hippel-Lindau disease.
* History of severe hypersensitivity to milk protein.
* Current use of any medication with strong anticholinergic properties, such as antihistamines, sleep aids, and antidiarrheal medications.
* Current use of indomethacin.
* Conditions that may result in low levels of releasable glucose in the liver and an inadequate reversal of hypoglycemia by glucagon such as prolonged fasting, starvation or chronic hypoglycemia as determined by the investigator.
* A positive response to any of the questions from the Physical Activity Readiness Questionnaire.
* Any chest discomfort with physical activity, including pain or pressure, or other types of discomfort.
* Any clinically significant disease or disorder which in the opinion of the Investigator may jeopardize the subject's safety or compliance with the protocol.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Castle, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Castle JR, El Youssef J, Wilson LM, Reddy R, Resalat N, Branigan D, Ramsey K, Leitschuh J, Rajhbeharrysingh U, Senf B, Sugerman SM, Gabo V, Jacobs PG. Randomized Outpatient Trial of Single- and Dual-Hormone Closed-Loop Systems That Adapt to Exercise Using Wearable Sensors. Diabetes Care. 2018 Jul;41(7):1471-1477. doi: 10.2337/dc18-0228. Epub 2018 May 11. PMID 29752345

RESULTS

PARTICIPANT FLOW:
Groups:
- SAP, PLGS, DH, SH: The randomization order for subjects in this arm was open loop (Sensor Augmented Pump SAP), predictive low glucose suspend (PLGS), dual hormone (DH) and single hormone (SH). Each visit was 84 hours and included inpatient and outpatient portions.
- SAP, DH, SH, PLGS: The randomization order for subjects in this arm was open loop (Sensor Augmented Pump SAP), dual hormone (DH), single hormone (SH) and predictive low glucose suspend (PLGS). Each visit was 84 hours and included inpatient and outpatient portions.
- DH, SH, SAP, PLGS: The randomization order for subjects in this arm was dual hormone (DH), single hormone (SH), open loop (Sensor Augmented Pump SAP), and predictive low glucose suspend (PLGS). Each visit was 84 hours and included inpatient and outpatient portions.
- SH, SAP, PLGS, DH: The randomization order for subjects in this arm was single hormone (SH), open loop (Sensor Augmented Pump SAP), predictive low glucose suspend (PLGS) and dual hormone (DH). Each visit was 84 hours and included inpatient and outpatient portions.
- PLGS, DH, SH, SAP: The randomization order for subjects in this arm was predictive low glucose suspend (PLGS), dual hormone (DH), single hormone (SH), and open loop (Sensor Augmented Pump SAP). Each visit was 84 hours and included inpatient and outpatient portions.
- PLGS, SAP, SH, DH: The randomization order for subjects in this arm was predictive low glucose suspend (PLGS), open loop (Sensor Augmented Pump SAP), single hormone (SH), and dual hormone (DH). Each visit was 84 hours and included inpatient and outpatient portions.
- SAP, DH, PLGS, SH: The randomization order for subjects in this arm was open loop (Sensor Augmented Pump SAP), dual hormone (DH), predictive low glucose suspend (PLGS), and single hormone (SH). Each visit was 84 hours and included inpatient and outpatient portions.
Period: Tslim Training Visit (2 Weeks)
Arm/Group | SAP, PLGS, DH, SH | SAP, DH, SH, PLGS | DH, SH, SAP, PLGS | SH, SAP, PLGS, DH | PLGS, DH, SH, SAP | PLGS, SAP, SH, DH | SAP, DH, PLGS, SH
Started | 4 | 1 | 8 | 5 | 5 | 1 | 1
Completed | 4 | 1 | 7 | 5 | 5 | 1 | 1
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: First Rest Period (1-12 Weeks)
Arm/Group | SAP, PLGS, DH, SH | SAP, DH, SH, PLGS | DH, SH, SAP, PLGS | SH, SAP, PLGS, DH | PLGS, DH, SH, SAP | PLGS, SAP, SH, DH | SAP, DH, PLGS, SH
Started | 4 | 1 | 7 | 5 | 5 | 1 | 1
Completed | 4 | 1 | 7 | 5 | 5 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: First Intervention (84 Hours)
Arm/Group | SAP, PLGS, DH, SH | SAP, DH, SH, PLGS | DH, SH, SAP, PLGS | SH, SAP, PLGS, DH | PLGS, DH, SH, SAP | PLGS, SAP, SH, DH | SAP, DH, PLGS, SH
Started | 4 | 1 | 7 | 5 | 5 | 1 | 1
Completed | 4 | 1 | 7 | 5 | 5 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Rest Period (7-45 Days)
Arm/Group | SAP, PLGS, DH, SH | SAP, DH, SH, PLGS | DH, SH, SAP, PLGS | SH, SAP, PLGS, DH | PLGS, DH, SH, SAP | PLGS, SAP, SH, DH | SAP, DH, PLGS, SH
Started | 4 | 1 | 7 | 5 | 5 | 1 | 1
Completed | 4 | 1 | 7 | 5 | 5 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (84 Hours)
Arm/Group | SAP, PLGS, DH, SH | SAP, DH, SH, PLGS | DH, SH, SAP, PLGS | SH, SAP, PLGS, DH | PLGS, DH, SH, SAP | PLGS, SAP, SH, DH | SAP, DH, PLGS, SH
Started | 4 | 1 | 7 | 5 | 5 | 1 | 1
Completed | 3 | 1 | 7 | 5 | 5 | 1 | 1
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Rest Period (7-45 Days)
Arm/Group | SAP, PLGS, DH, SH | SAP, DH, SH, PLGS | DH, SH, SAP, PLGS | SH, SAP, PLGS, DH | PLGS, DH, SH, SAP | PLGS, SAP, SH, DH | SAP, DH, PLGS, SH
Started | 3 | 1 | 7 | 5 | 5 | 1 | 1
Completed | 3 | 1 | 6 | 5 | 4 | 1 | 1
Not Completed | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1 | 0 | 0
Period: Third Intervention (84 Hours)
Arm/Group | SAP, PLGS, DH, SH | SAP, DH, SH, PLGS | DH, SH, SAP, PLGS | SH, SAP, PLGS, DH | PLGS, DH, SH, SAP | PLGS, SAP, SH, DH | SAP, DH, PLGS, SH
Started | 3 | 1 | 6 | 5 | 4 | 1 | 1
Completed | 3 | 1 | 6 | 4 | 4 | 1 | 1
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — diagnosis of gastroparesis | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Fourth Rest Period (7-45 Days)
Arm/Group | SAP, PLGS, DH, SH | SAP, DH, SH, PLGS | DH, SH, SAP, PLGS | SH, SAP, PLGS, DH | PLGS, DH, SH, SAP | PLGS, SAP, SH, DH | SAP, DH, PLGS, SH
Started | 3 | 1 | 6 | 4 | 4 | 1 | 1
Completed | 3 | 1 | 6 | 4 | 4 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Fourth Intervention (84 Hours)
Arm/Group | SAP, PLGS, DH, SH | SAP, DH, SH, PLGS | DH, SH, SAP, PLGS | SH, SAP, PLGS, DH | PLGS, DH, SH, SAP | PLGS, SAP, SH, DH | SAP, DH, PLGS, SH
Started | 3 | 1 | 6 | 4 | 4 | 1 | 1
Completed | 3 | 1 | 6 | 4 | 4 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Type 1 diabetics using an insulin pump
Groups:
- All Study Participants: All study participants were randomized to complete four 84 hour study visits using either standard of care insulin pump therapy, dual hormone, single hormone or predictive low glucose suspend closed loop control. Treatment order was randomized.
Arm/Group | All Study Participants
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Percent of Time With Sensed Glucose < 3.9 mmol/L
Description: Assess the percent of time that the Dexcom G4 Share reported sensor glucose values less than 3.9 mmol/L using Dexcom sensor downloads across all four arms.
Time Frame: entire 84 hour study
Population: All subjects analyzed for those who started a PLGS, SH, DH or SAP arm.
Measure: Mean (Standard Deviation); unit: percentage of 84 hours
Groups:
- Predictive Low Glucose Suspend Arm: The predictive low glucose suspend system will run through the artificial pancreas controller in predictive low glucose suspend mode and utilize the patient's optimized basal rates, correction factor, and carb ratio, but it will have the additional safety net of the pump suspending insulin when it predicts a hypoglycemic event.
  Artificial Pancreas Controller in Predictive Low Glucose Suspend Mode: The artificial pancreas controller contains an algorithm for managing blood glucose in people with type 1 diabetes which includes an exercise detection component. The new algorithm will have 3 modes: a single hormone closed-loop insulin only mode, a dual-hormone closed-loop insulin and glucagon mode and an insulin only mode with predictive low glucose suspend. Closed-loop Artificial Pancreas Controller includes insulin delivery algorithm implemented on a smart phone, utilizing sensor glucose values from a Dexcom G4 sensor and sending delivery command
- Dual Hormone Closed-loop Arm: Artificial Pancreas Controller in Dual Hormone Mode: The artificial pancreas controller contains an algorithm for managing blood glucose in people with type 1 diabetes which includes an exercise detection component. The new algorithm will have 3 modes: a single hormone closed-loop insulin only mode, a dual-hormone closed-loop insulin and glucagon mode and an insulin only mode with predictive low glucose suspend. Closed-loop Artificial Pancreas Controller includes insulin and glucagon delivery algorithm implemented on a smart phone, utilizing sensor glucose values from a Dexcom G4 sensor and sending delivery commands to two Tandem t:slim insulin pumps, one filled
Arm/Group | Predictive Low Glucose Suspend Arm | Dual Hormone Closed-loop Arm | Single Hormone Closed-loop Arm | Sensor Augmented Pump Therapy Arm
Number analyzed (Participants) | 23 | 22 | 22 | 22
percentage of 84 hours | 1.8 (1.5) | 1.2 (1.0) | 2.7 (1.7) | 3.0 (3.1)

2. Primary Outcome: Percent of Time With Sensed Glucose < 3.9 mmol/L
Description: as for outcome 1
Time Frame: From 14:00-18:00 for each 12 hour inpatient visit
Population: All subjects analyzed for those who started a PLGS, SH, DH or SAP arm.
Measure: Mean (Standard Deviation); unit: percentage of 4 hours after exercise
Arm/Group | Predictive Low Glucose Suspend Arm | Dual Hormone Closed-loop Arm | Single Hormone Closed-loop Arm | Sensor Augmented Pump Therapy Arm
Number analyzed (Participants) | 23 | 22 | 22 | 22
percentage of 4 hours after exercise | 6.9 (8.0) | 3.5 (4.9) | 7.5 (12.2) | 4.0 (6.6)

3. Primary Outcome: Percent of Time With Sensed Glucose Between 3.9-10 mmol/L
Description: Assess the percent of time that the Dexcom G4 Share reported sensor glucose values between 3.9-10 mmol/L using Dexcom sensor downloads across all four arms.
Time Frame: entire 84 hour study
Population: All subjects analyzed for those who started a PLGS, SH, DH or SAP arm.
Measure: Mean (Standard Deviation); unit: percentage of 84 hours
Arm/Group | Predictive Low Glucose Suspend Arm | Dual Hormone Closed-loop Arm | Single Hormone Closed-loop Arm | Sensor Augmented Pump Therapy Arm
Number analyzed (Participants) | 23 | 22 | 22 | 22
percentage of 84 hours | 62.9 (14.5) | 72.7 (10.5) | 75.6 (8.7) | 63.1 (17.6)

4. Primary Outcome: Percent of Time With Sensed Glucose Between 3.9-10 mmol/L
Description: as for outcome 3
Time Frame: From 14:00-18:00 for each 12 hour inpatient visit
Population: All subjects analyzed for those who started a PLGS, SH, DH or SAP arm.
Measure: Mean (Standard Deviation); unit: percentage of 4 hours after exercise
Arm/Group | Predictive Low Glucose Suspend Arm | Dual Hormone Closed-loop Arm | Single Hormone Closed-loop Arm | Sensor Augmented Pump Therapy Arm
Number analyzed (Participants) | 23 | 22 | 22 | 22
percentage of 4 hours after exercise | 78.0 (20.1) | 84.6 (16.1) | 84.4 (16.3) | 79.4 (25.3)

5. Secondary Outcome: Mean Sensed Glucose
Description: Assess the mean sensor glucose using Dexcom sensor downloads across all four arms.
Time Frame: entire 84 hour study
Population: All subjects analyzed for those who started a PLGS, SH, DH or SAP arm.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Predictive Low Glucose Suspend Arm | Dual Hormone Closed-loop Arm | Single Hormone Closed-loop Arm | Sensor Augmented Pump Therapy Arm
Number analyzed (Participants) | 23 | 22 | 22 | 22
mg/dL | 165.9 (21.8) | 154.1 (15.8) | 146.8 (12) | 161.9 (29)

6. Secondary Outcome: Number of Carbohydrate Treatments
Description: Assess the number of rescue carbohydrate treatments per day across all four arms.
Time Frame: entire 84 hour study
Population: All subjects analyzed for those who started a PLGS, SH, DH or SAP arm.
Measure: Mean (Standard Deviation); unit: number of carbohydrate treatments/day
Arm/Group | Predictive Low Glucose Suspend Arm | Dual Hormone Closed-loop Arm | Single Hormone Closed-loop Arm | Sensor Augmented Pump Therapy Arm
Number analyzed (Participants) | 23 | 22 | 22 | 22
number of carbohydrate treatments/day | 1.3 (1.3) | 0.8 (0.7) | 1.6 (1.4) | 1.4 (1.2)

7. Secondary Outcome: Percent of Time With Sensed Glucose < 3.0 mmol/L
Description: Assess the percent of time that the Dexcom G4 Share reported sensor glucose values less than 3.0 mmol/L using Dexcom sensor downloads across all four arms.
Time Frame: entire 84 hour study
Population: All subjects analyzed for those who started a PLGS, SH, DH or SAP arm.
Measure: Mean (Standard Deviation); unit: percentage of 84 hours
Arm/Group | Predictive Low Glucose Suspend Arm | Dual Hormone Closed-loop Arm | Single Hormone Closed-loop Arm | Sensor Augmented Pump Therapy Arm
Number analyzed (Participants) | 23 | 22 | 22 | 22
percentage of 84 hours | 0.2 (0.3) | 0.2 (0.4) | 0.6 (0.6) | 0.3 (0.6)

8. Secondary Outcome: Percent of Time With Sensed Glucose > 10 mmol/L
Description: Assess the percent of time that the Dexcom G4 Share reported sensor glucose values greater than 10 mmol/L using Dexcom sensor downloads across all four arms
Time Frame: entire 84 hour study
Population: All subjects analyzed for those who started a PLGS, SH, DH or SAP arm.
Measure: Mean (Standard Deviation); unit: percentage of 84 hours
Arm/Group | Predictive Low Glucose Suspend Arm | Dual Hormone Closed-loop Arm | Single Hormone Closed-loop Arm | Sensor Augmented Pump Therapy Arm
Number analyzed (Participants) | 23 | 22 | 22 | 22
percentage of 84 hours | 35.2 (15.1) | 26.1 (10.9) | 21.7 (9.1) | 33.9 (18.2)

9. Secondary Outcome: Number of Events With Capillary Blood Glucose < 3.9 mmol/L
Description: Assess number of events with capillary blood glucose < 3.9 mmol/L using downloads from a Contour Next blood glucose meter across all four arms. .
Time Frame: entire 84 hour study
Population: All subjects analyzed for those who started a PLGS, SH, DH or SAP arm.
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | Predictive Low Glucose Suspend Arm | Dual Hormone Closed-loop Arm | Single Hormone Closed-loop Arm | Sensor Augmented Pump Therapy Arm
Number analyzed (Participants) | 23 | 22 | 22 | 22
number of events | 0.8 (0.7) | 0.7 (0.5) | 1.1 (0.7) | 0.9 (0.9)

10. Secondary Outcome: Number of Events With Capillary Blood Glucose < 3.0 mmol/L
Description: Assess number of events with capillary blood glucose < 3.0 mmol/L using downloads from a Contour Next blood glucose meter across all four arms.
Time Frame: entire 84 hour study
Population: All subjects analyzed for those who started a PLGS, SH, DH or SAP arm.
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | Predictive Low Glucose Suspend Arm | Dual Hormone Closed-loop Arm | Single Hormone Closed-loop Arm | Sensor Augmented Pump Therapy Arm
Number analyzed (Participants) | 23 | 22 | 22 | 22
number of events | 0.1 (0.1) | 0.1 (0.2) | 0.2 (0.3) | 0.1 (0.2)

11. Secondary Outcome: Mean Amount of Insulin Delivered
Description: Assess the average amount of insulin delivered per day in units/kg as documented through the artificial pancreas controller across all four arms.
Time Frame: 24 hours
Population: All subjects analyzed for those who started a PLGS, SH, DH or SAP arm.
Measure: Mean (Standard Deviation); unit: units/kg
Arm/Group | Predictive Low Glucose Suspend Arm | Dual Hormone Closed-loop Arm | Single Hormone Closed-loop Arm | Sensor Augmented Pump Therapy Arm
Number analyzed (Participants) | 23 | 22 | 22 | 22
units/kg | 43.8 (17.5) | 44.2 (16.0) | 42.6 (14.1) | 44.1 (13.2)

12. Secondary Outcome: Mean Amount of Glucagon Delivered
Description: Assess the average amount of insulin delivered per day in units/kg as documented through the artificial pancreas controller in dual hormone arm.
Time Frame: 24 hours
Population: All subjects analyzed for those who started a PLGS, SH, DH or SAP arm.
Measure: Mean (Standard Deviation); unit: mcg/kg
Groups:
- Dual Hormone Closed Loop: Artificial Pancreas Controller in Dual Hormone Mode: The artificial pancreas controller contains an algorithm for managing blood glucose in people with type 1 diabetes which includes an exercise detection component. The new algorithm will have 3 modes: a single hormone closed-loop insulin only mode, a dual-hormone closed-loop insulin and glucagon mode and an insulin only mode with predictive low glucose suspend. Closed-loop Artificial Pancreas Controller includes insulin and glucagon delivery algorithm implemented on a smart phone, utilizing sensor glucose values from a Dexcom G4 sensor and sending delivery commands to two Tandem t:slim insulin pumps, one filled with insulin and one with glucagon
Arm/Group | Dual Hormone Closed Loop | Predictive Low Glucose Suspend Arm | Single Hormone Closed-loop Arm | Sensor Augmented Pump Therapy Arm
Number analyzed (Participants) | 23 | 22 | 22 | 22
mcg/kg | 516.1 (201.1) | 0 (0) | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: 12 months
Description: All participants that began/started the tslim training visit or a PLGS, SH, DH or SAP arm are included in the adverse events. The numbers from the participant flow indicate 25 subjects began the tslim training visit, 23 subjects began a PLGS visit, and 22 subjects began a DH, SH or SAP visit.
Groups:
- Tslim Training: Subjects used the tslim and Dexcom G4 Share of G5 sensor for two weeks at home to allow subjects to become familiar with the devices.
Arm/Group | Predictive Low Glucose Suspend Arm | Dual Hormone Closed-loop Arm | Single Hormone Closed-loop Arm | Sensor Augmented Pump Therapy Arm | Tslim Training
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22 | 0/22 | 0/22 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22 | 0/22 | 0/22 | 0/25
Other Adverse Events (participants affected / at risk) | 5/23 | 8/22 | 2/22 | 3/22 | 2/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Predictive Low Glucose Suspend Arm (N=23) | Dual Hormone Closed-loop Arm (N=22) | Single Hormone Closed-loop Arm (N=22) | Sensor Augmented Pump Therapy Arm (N=22) | Tslim Training (N=25)
GI upset (Gastrointestinal disorders) | 3 (6) | 4 (8) | 0 (0) | 1 (1) | 0 (0) — GI upset includes: nausea, stomach cramps, belching, sour stomach.
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
mild edema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — minor pain and redness at IV or infusion site
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) — Rash at a sensor insertion site or from heart rate monitor.
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
device induced symptomatic hypoglycemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lightheadedness (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT02862730/Prot_SAP_000.pdf